CLINICAL TRIAL: NCT03105284
Title: Adipose-tissue Derived Stem Cells: Characterization of Adipose-tissue Derived Stem Cells in Flaps Versus Liposuction
Brief Title: Adipose-tissue Derived Stem Cells in Flaps Versus Liposuction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ASC Aarhus
Record Dates: First submitted 2017-02-27; First posted 2017-04-07 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-02

CONDITIONS: Mesenchymal Stem Cells
Keywords: stem cell; liposuction; regenerative medicine
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Intervention Model Description: Participants will act as their own control. Each participant will receive both excision and liposuction of fat.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposuction of fat (Active Comparator): The intervention examined is the extraction method by liposuction.
  Interventions: Procedure: Liposuction
- Excision of fat (No Intervention): Control group

INTERVENTIONS:
Procedure: Liposuction — Fat harvest by liposuction (Colemans method)
  Arms: Liposuction of fat

SUMMARY:
The aim of the study is to evaluate a physiological concentration of adipose tissue-derived stem cells (ASC) in excised fat versus fat harvested by liposuction. Participants will act as their own control as both extraction methods are performed on each participant.

DETAILED DESCRIPTION:
Adipose tissue-derived stem cells are of great interest due to their relevance in regenerative medicine and tissue engineering. A reason, being their capacity for multipotent differentiation, tissue repair and immune modulation.

To evaluate a physiological concentration level of ASCs in human fat we investigate two extraction methods of fat, excision and liposuction. This is done through a standardised setup with patients acting their own control. The study is carried out in accordance with the guidelines provided by the International Federation for Adipose Therapeutics and Science and International Society for Cellular Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women - over the age of 18
* Deemed suitable for abdominoplasty with abdomen pendens, fleur de lis, panniculectomy or belt lipectomy.
* Able to read and understand Danish

Exclusion Criteria:

* Current smokers - patients not having paused for a minimum of four weeks prior to surgery.
* Prior or current adjuvant chemo therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Stem cell yield | At baseline right after isolation.
  Stem cell yield measured by antibody stained flow cytometry.
Stem cell yield | Cells are cultured from baseline to day 14.
  Stem cell yield measured by colony forming units and number of colonies >50 cells are counted.

SECONDARY OUTCOMES:
Growth kinetics | Cultured for 7 days and counted.
  Growth kinetics measured by culturing. The population doubling time is determined using log phase of growth
Adipogenic, chondrogenic and osteogenic differentiation. | Through study completion, an average of 1 year.
  Differentiation assays for adipogenic, chondrogenic and osteogenic differentiation with Oil Red O staining, Safranin O staining and Alizarin red S staining.

REFERENCES:
- [Background] Bourin P, Bunnell BA, Casteilla L, Dominici M, Katz AJ, March KL, Redl H, Rubin JP, Yoshimura K, Gimble JM. Stromal cells from the adipose tissue-derived stromal vascular fraction and culture expanded adipose tissue-derived stromal/stem cells: a joint statement of the International Federation for Adipose Therapeutics and Science (IFATS) and the International Society for Cellular Therapy (ISCT). Cytotherapy. 2013 Jun;15(6):641-8. doi: 10.1016/j.jcyt.2013.02.006. Epub 2013 Apr 6. PMID 23570660
- [Derived] Alstrup T, Eijken M, Brunbjerg ME, Hammer-Hansen N, Moller BK, Damsgaard TE. Measured Levels of Human Adipose Tissue-Derived Stem Cells in Adipose Tissue Is Strongly Dependent on Harvesting Method and Stem Cell Isolation Technique. Plast Reconstr Surg. 2020 Jan;145(1):142-150. doi: 10.1097/PRS.0000000000006404. PMID 31881616